CLINICAL TRIAL: NCT06898489
Title: Traditional Chinese Five-Tone Therapy As an Adjunctive Treatment for Systemic Lupus Erythematosus: a Prospective Cohort Study
Brief Title: Adjunctive Yu-Tone Music Therapy for Systemic Lupus Erythematosus: a Prospective Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: Yijun Luo (Other Government)
Responsible Party: Sponsor-Investigator, Yijun Luo, PhD Candidate, Zhejiang Chinese Medical University
Organization: Zhejiang Chinese Medical University (Other Government)
Other Study IDs: 20250228-3
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Systemic Lupus Erythematosus; Music Therapy
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control group: No Yu-tone music intervention, receiving conventional pharmacotherapy only.
  Interventions: Drug: Conventional pharmacotherapy
- Yu-Tone Music Intervention Group: In addition to conventional pharmacotherapy, SLE patients receive a structured Yu-tone music listening program
  Interventions: Combination Product: Yu-Tone Music Intervention; Drug: Conventional pharmacotherapy

INTERVENTIONS:
Combination Product: Yu-Tone Music Intervention — SLE patients undergo a structured Yu-tone music listening program (30 minutes daily, 5 days per week, with each cycle lasting 8 weeks, for a total of 3 cycles
  Groups: Yu-Tone Music Intervention Group
Drug: Conventional pharmacotherapy — Standard SLE medications (e.g., hydroxychloroquine, glucocorticoids).

SUMMARY:
The goal of this observational study is to investigate the long-term adjunctive effects of Traditional Chinese Five-Tone Therapy (Yu Tone) in patients with systemic lupus erythematosus (SLE). The main question it aims to answer is:

Does Yu-tone music therapy improve psychological well-being and quality of life in SLE patients when used as a complementary intervention alongside standard pharmacotherapy? Participants already receiving Yu-tone music therapy as part of their integrative care for SLE will complete validated online questionnaires assessing psychological distress (e.g., anxiety, depression), disease-related quality of life, and medication adherence monthly for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Meet the 2019 ACR/EULAR classification criteria for SLE; ② Adults aged 18 years or older; ③ Provide informed consent to participate in the study.

Exclusion Criteria:

* Presence of severe organ dysfunction (e.g., renal failure, cardiac insufficiency) or psychiatric disorders; ② Diagnosed with hearing impairment or auditory disorders; ③ Inability to comprehend or complete study questionnaires (e.g., due to cognitive impairment or language barriers).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study Population are Chinese
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
SLEDAI score | From enrollment to the treatment at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou, 310053, China., Hangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided